CLINICAL TRIAL: NCT01730430
Title: Investigation of Biomarkers of Disease State in Alzheimer's Disease and Non-AD Dementias
Brief Title: Cerebrospinal Fluid (CSF) Biomarkers Alzheimer's Disease (AD) and Non-AD Dementias
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: Pro00033660
Record Dates: First submitted 2012-10-17; First posted 2012-11-21 (Estimated); Last update posted 2014-04-22 (Estimated); Status verified 2014-04

CONDITIONS: Alzheimer's Disease; Dementias
Keywords: non-AD dementias; healthy elderly controls
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood, urine and cerebral spinal fluid.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Collection of CSF: 1. Those with Alzheimer's disease
  2. Those with non-Alzheimer's disease dementia
  3. Healthy elderly volunteers

SUMMARY:
To establish a cutoff value using a ratio of CSF tau to Aβ42 (tau/Aβ42) for distinguishing patients wth mild to moderate Alzheimer's disease (AD) from health elderly control subjects. The investigators hypothesize that a cutoff can be found that has at least 80% sensitivity and 60% specificity.

DETAILED DESCRIPTION:
This study will enroll 50 AD subjects, 50 normal controls and approximately 20 subjects with non-AD dementia. There will be 2 visits (up to 30 days apart), and a telephone follow-up visit.

This protocol does not include treatment of subjects. Lumbar puncture and phlebotomy are routine clinical tasks and are associated with a low level of risk. All adverse events will be documented and reviewed by the PI.

ELIGIBILITY:
Inclusion Criteria:

* Each subject must be ≥ 55 to ≤ 85 years of age.
* Each subject must be able to read at a 6th grade level, as determined by the investigator, and must have a history of academic achievement and/or employment sufficient to exclude mental retardation.
* Each subject must have results of clinical laboratory tests, a physical examination, vital signs within normal limits or clinically acceptable to the investigator within 28 days prior to enrollment.
* Each subject (or legal representative) must sign the informed consent form after the scope and nature of the investigation have been explained to them, and before screening assessments.

Additional Inclusion Criteria for Normal Controls:

* Must have a global Clinical Dementia Rating (CDR) score of 0.
* Must have a Mini-Mental State Examination (MMSE) score ≥ 28.
* Must have a Z-score ≥ -1.0 in each cognitive domain of memory (including delayed recall), language, executive function and attention, and visuoconstruction with neuropsychological tests of choice and adjustment for age, gender, and education level if indicated.

Additional Inclusion Criteria for AD Subjects:

* Must meet the criteria for a diagnosis of probable AD based on both

  1. the National Institute of Neurological and Communicative Diseases and Stroke/Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria, and
  2. the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition, Text Revision (DSM IV TR) criteria for AD.
* Must have an MMSE score ≥ 15 and ≤ 26.
* Must have a clear history of cognitive and functional decline over at least one year that is either

  1. documented in medical records or
  2. documented by history from an informant who knows the subject well.
* Must have an MRI or CT scan that is consistent with a diagnosis of AD within 12 months prior to enrollment.

Exclusion Criteria for AD Subjects and Normal Controls

* The subject has a Rosen modified Hachinski Ischemia Score > 4.
* The subject has a known history of stroke.
* The subject has evidence of a clinically relevant or unstable neurological or psychiatric disorder (for AD subjects - other than AD).
* The subject has a history of alcoholism or drug dependency/abuse within the last 5 years before enrollment.
* The subject has an ongoing uncontrolled, clinically significant medical condition such that, in the judgment of the investigator, a subject's participation in the trial would pose a significant medical risk to the subject.
* The subject has participated within the last two months in a clinical trial of a novel therapeutic agent (e.g. bapineuzumab) or has ever been in a clinical trial of an AD vaccine.
* Pregnancy

Additional Inclusion and Exclusion Criteria for Subject with non-AD dementias

* Standard clinical diagnostic criteria accepted by the field for non-AD dementias should be used by the Institution.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Duke Memory Disorders Clinic
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2012-07; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Ratio of CSF tau to Aβ42 (tau/Aβ42) | CSF will be collected at Visit 1 (up to 30 days after the screening visit)
  CSF will be collected in clinic and shipped frozen to Merck's Clinical Development Lab for testing. Any remaining samples will be kept up to 20 years.

CONTACTS AND LOCATIONS:
Overall Officials: James Burke, MD, PhD, Principal Investigator — Duke UMC
Locations (1):
- Duke Health Center at Morreene Road, Durham, North Carolina, United States